CLINICAL TRIAL: NCT06958055
Title: Vallecular Bolus Aggregation During Swallowing of Solid Food Boluses for Subject Rehabilitated With Mandibular Implant Retained Overdentures. A Crossover Study
Brief Title: Vallecular Bolus Aggregation During Swallowing for Implant Overdenture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A0102025RP
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Prosthesis Durability
Keywords: vallecular aggregation; swallowing; solid food; implant overdenture
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group I : complete edentulous patients (Placebo Comparator): videofluroscopy for completely edentulous patients
  Interventions: Radiation: videofluroscopy evaluation of swallowing function
- group II: Conventional complete denture (Active Comparator): complete denture construction for edentulous patient and videofluroscopy evaluation
  Interventions: Radiation: videofluroscopy evaluation of swallowing function
- group III: Implant overdentutres (Active Comparator): construction of implant overdenture and videofluroscopy evaluation
  Interventions: Radiation: videofluroscopy evaluation of swallowing function

INTERVENTIONS:
Radiation: videofluroscopy evaluation of swallowing function — Videofluoroscopy swallowing evaluation was done using solid food bolus at three different oral conditions: Without dentures (WOD), with the conventional complete denture (CDs) and with mandibular implant retained overdenture (IODs).

SUMMARY:
evaluate the effect of implant retained mandibular overdenture on vallecular bolus aggregation during chewing and subsequent swallowing of solid food consistency.

DETAILED DESCRIPTION:
Healthy edentulous subjects seeking prosthetic treatment at the prosthodontics department, Faculty of Dentistry, Mansoura University will be eligible for this study. The inclusion criteria will be: age >60 year; Class I maxilla-mandibular relation; available inter-arch space; and adequate bone quality and quality in the mandibular anterior alveolar ridge (inter-foraminal area). Subjects with physical or cognitive limitations, neurodegenerative disorders that could influence their swallowing function, parafunctional habits, smokers, signs or symptoms of temporomandibular disorders, osteoporosis, uncontrolled systemic diseases, previously undergone radiotherapy or laryngeal surgery will be excluded from the study.

Sample size estimation is based on a previous study evaluated the oral and pharyngeal phases of swallowing by videofluroscopy and found significant differences between groups. We determined that 16 participants will be required for the detection of significant differences with effect size of 0.78, 90% power, and 5% error probability. Ethical agreement will be taken from ethical committee of the faculty of dentistry and written consent will be gotten from all the participants after illustrating in detail the whole research protocol.

Prosthetic and surgical procedures:

For each patient, new conventional complete denture will be constructed with optimal denture extension and lingualized balanced occlusal scheme. The new prosthesis will be inserted intraorally and adjusted for occlusal interferences. Subsequently, two dental implants will be placed in the canines region according to guided surgery protocol and two-stage approach. After osseointegration, locator attachments will be screwed to the dental implants to convert the conventional mandibular denture to mandibular implant retained overdenture. The mandibular implant overdentutre will be inserted and occlusal adjustment will be done and follow up visits will be scheduled.

II- Evaluation method:

Each patient will be subjected to videofluoroscopic imaging at 3 different oral conditions; without denture, after 3 months of complete dentures insertion, and after 3 months of mandibular implant overdenture insertion.

Videofluroscopic (VF) assessment:

All participants will be evaluated by using videofluoroscopic evaluation of bolus movement. Each patient will be asked to chew ¼ of cookie (coated with pudding and barium powder) and swallow the bolus once they will be ready. The videofluoroscopic recordings will be transferred to the computer for later data analysis. EO program (Version 1.36) was used to analyze the videofluoroscopic recordings by placing numbers (1/100 second) on the video frame for later frame-by-frame data analysis.

The following parameters will be measured:

* Bolus location at swallow onset (BLSO).
* Swallow reaction time (SRT), that is, the interval, from bolus passing the mandible (BPM) to hyoid burst (HYB) onset.
* Vallecular aggregation time (VAT), that is, the interval, from BPM to end of aggregation (EOA), with EOA defined as the first frame showing the leading edge of the bolus moving below the level of the pit of the vallecular space.
* The EOA-to-HYB interval.

ELIGIBILITY:
Inclusion Criteria:

* age >60 year.
* Class I maxilla-mandibular relation;
* Available inter-arch space.
* adequate bone quality and quality in the mandibular anterior alveolar ridge (inter-foraminal area).

Exclusion Criteria:

* Subjects with physical or cognitive limitations,
* Neurodegenerative disorders that could influence their swallowing function,
* Parafunctional habits,
* Smokers,
* Signs or symptoms of temporomandibular disorders,
* Osteoporosis,
* Uncontrolled systemic diseases,
* Previously undergone radiotherapy or laryngeal surgery

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
swallowing evaluation | after 3 months of denture and overdenture insertion
  videofluroscopy evaluation for swallowing function

CONTACTS AND LOCATIONS:
Overall Officials: abdallah M Ibrahim, PhD, Principal Investigator — Mansoura university, Faculty of dentistry, prosthodontics department
Locations (1):
- faculty of dentistry, mansoura university Mansoura, Egypt,, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ibrahim AM, Elgamal M, Abdel-Khalek EA. Hyoid displacement during swallowing function for completely edentulous subjects rehabilitated with mandibular implant retained overdenture. BMC Oral Health. 2024 Aug 8;24(1):914. doi: 10.1186/s12903-024-04616-9. PMID 39118020